CLINICAL TRIAL: NCT05129579
Title: The Effect of the Mindfulness Based Stress Reduction Intervention on Psychological Resilience and Psychological Well-being of Intensive Care Nurses
Brief Title: Psychological Resilience and Psychological Well-being of Intensive Care Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Responsible Party: Principal Investigator, Merve BAT TONKUŞ, Lecturer, PhD Cand., İstanbul Yeni Yüzyıl Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulYeniYU
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Psychological Resilience; Well-being
Keywords: Mindfulness; Intensive Care Nurses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBRSEG (Experimental): The group in which the mindfulness-based stress reduction intervention will be implemented.
  Interventions: Behavioral: Mindfulness Based Stress Reduction Intervention
- control group (Other): The group to which mindfulness-based stress reduction intervention will not be applied
  Interventions: Other: no intervention

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Intervention — Mindfulness Based Stress Reduction intervention is a manualized course that includes meditation, relaxing movement, and breathing. A certified MBSR instructor will teach the courses in a group-based format for 90 minute sessions, once per week for eight weeks.
  Arms: MBRSEG
Other: no intervention — No intervention will be made in the control group.
  Arms: control group

SUMMARY:
Purpose: This study aims to determine the impact of mindfulness-based stress reduction programs on the psychological resilience and well-being of intensive care nurses.

Design: The study was planned as an experimental study with a randomized control group, using pre-test, post-test and follow-up test.

Hypotheses: H1: The resilience level scores of the nurses in the intervention group participating in the mindfulness-based stress reduction initiative will increase compared to the nurses in the control group.

H2: Nurses in the intervention group participating in the mindfulness-based stress reduction initiative will increase their well-being level scores compared to the nurses in the control group.

H3: The psychological resilience level posttest and follow-up scores of the nurses in the intervention group participating in the mindfulness-based stress reduction initiative will increase compared to their pretest scores.

H4: The well-being level posttest and follow-up scores of the nurses in the intervention group participating in the mindfulness-based stress reduction initiative will increase according to their pretest scores.

ELIGIBILITY:
Inclusion Criteria:

* Having Having a working time of at least 6 months in the intensive care unit,
* No barriers to accessing technology for participation in the online training program,
* Absence of a communication barrier related to vision and hearing

Exclusion Criteria:

* Working in the intensive care unit for less than 6 months
* Working in the intensive care unit due to temporary assignment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Psychological Resilience Level | for 3 months
  Psychological Resilience Scale for Adults: The scale consists of 33 items; it includes 6 sub-dimensions: The structural style (3,9,15,21) and perception of future (2,8,14,20) subdimensions were measured by 4 items each, the family cohesion (5,11,17,23,26,32), perception of self (1,7,13,19,28,31,), and social competence (4,10,16,22,25,29) sub-dimensions were measured by 6 items each, and the social resources (6,12,18,24,27,30,33) sub-dimension was measured by 7 items. The score that can be obtained from the scale varies from 33 to 165.
Psychological Well-being Level | for 3 months
  Psychological Well-Being Scale: The items of the scale are answered between 1 and 7, as I strongly disagree (1) and I strongly agree (7). All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items). A high score indicates that the person has many psychological resources and strengths.

IPD SHARING:
Plan to Share IPD: No